CLINICAL TRIAL: NCT05316662
Title: A Multi-centre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Use of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in Mexico
Brief Title: A Research Study Looking at How Oral Semaglutide Works in People With Type 2 Diabetes in Mexico, as Part of Local Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4645; U1111-1240-4396 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semaglutide: Participants with T2D will be assessed for clinical parameters associated with the once-daily use of oral semaglutide who have not previously been treated with injectable glucose-lowering medication in routine clinical practice.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the participant in this study.

SUMMARY:
The purpose of the study is to collect information on how Rybelsus® works in people with type 2 diabetes and to see if Rybelsus® can lower participant's blood sugar levels. Participants will get Rybelsus® as prescribed by the study doctor. The study will last for about 8-10 months. Participant will be asked to complete a questionnaire about how the participant will take Rybelsus® tablets. Participant will complete this questionnaire during the normally scheduled visit with the study doctor. Participant will be asked to complete some questionnaires about diabetes treatment. Participant will complete these questionnaires during normally scheduled visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Diagnosed with type 2 diabetes mellitus
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Available HbA1c value less than or equal to 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (V1) if in line with local clinical practice
* Treatment naive to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than 14 days

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Treatment with any investigational drug within 30 days prior to enrolment into the study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with T2D will be assessed for clinical parameters associated with the once-daily use of oral semaglutide who have not previously been treated with injectable glucose-lowering medication in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in percentage (%)-points

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in percentage (%)
Absolute change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in Kilogram (Kg)
HbA1c < 7% | End of Study visit (V3) (week 34- 44)
  Measured as Yes or No
HbA1c reduction >=1%-points and body weight reduction of >=5% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No
HbA1c reduction >=1%-points and body weight reduction of >=3% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No
DTSQc, relative treatment satisfaction | End of Study visit (V3) (week 34- 44)
  Measured in Total score
DTSQs, change in absolute treatment satisfaction | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in Total score

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- Mexico (2):
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - CICEJ Centro de Investigacion Clinica Endocrinologica de Jalisco SC, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com